CLINICAL TRIAL: NCT05023265
Title: Assessment of Quality of Life and Outcomes in Patients Treated With Stereotactic Body Radiotherapy (SBRT) for Inoperable Renal Cell Carcinoma (RCC): A Multicenter Phase II Study
Brief Title: Assessment of Quality of Life and Outcomes in Patients With Primary Renal Cell Carcinoma Treated With SBRT
Acronym: AQuOS-II
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Juravinski Cancer Center (Other); St. Joseph's Healthcare Hamilton (Other); The Ottawa Hospital (Other); Health Sciences North (Other); Grand River Regional Cancer Centre (Other); British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Dr. William Chu, Assistant Professor, Dept of Radiation Oncology Sunnybrook Odette Cancer Centre, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3641
Record Dates: First submitted 2021-08-05; First posted 2021-08-26 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with Inoperable Renal Cell Carcinoma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT for Medically Inoperable RCC (Experimental): 35-40 Gy in five fractions (7-8 Gy/day)
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — SBRT is a non-invasive treatment approach that delivers precise and highly conformal radiotherapy to the tumour with steep dose gradients that minimize exposure to the surrounding normal tissues.

SUMMARY:
This is a multicenter, single arm phase II study of stereotactic body radiation therapy (SBRT) for patients with medically inoperable primary renal cell carcinoma (RCC).

DETAILED DESCRIPTION:
Primary renal cell carcinoma (RCC) is a common malignancy in Canada. The current standard of care for fit patients with localized RCC is surgical resection of the kidney (nephrectomy). RCC, however, affects predominately an older population with a median age at diagnosis of 65 years. Surgery is often not an option for these patients due to existing co-morbidities, and in an increasing environment of shared decision making in healthcare, some patients decline surgical resection and seek less invasive alternatives.

Stereotactic body radiotherapy (SBRT) is a treatment approach that offers precise delivery of highly conformal radiotherapy to the tumour with minimal exposure to the surrounding normal tissues. SBRT is non-invasive and not limited by the size or location of kidney tumors like other ablative strategies. The worldwide experience of treating RCC with SBRT is growing and the results to date are promising. There is broader enthusiasm from both the radiation oncology and urology community to increase utilization of SBRT for RCC in non-surgical patients within the context of a well-designed prospective trial in Canada.

We will prospectively assess the efficacy, toxicity and impact on quality of life (QoL) of SBRT in the treatment of inoperable RCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years old
* Newly diagnosed RCC by biopsy (preferred) or radiologic evidence of growth on surveillance over two consecutive assessments (6-12 months)
* Primary lesion >3 cm, or recurrent lesion following local ablative therapy
* Medically inoperable or patient who refuses surgery following assessment by experienced urologist, and discussed in a multidisciplinary setting
* ECOG 0-2
* Written informed consent
* Participants must be able to understand the English-language or with the aid of a translator

Exclusion Criteria:

* Primary Lesion >20cm
* Evidence of distant metastatic disease
* Previous abdominal RT in vicinity of kidney preventing definitive SBRT
* History of major radiosensitivity syndrome
* Second invasive malignancy within the past 3 years (excluding non-melanomatous skin cancer)
* Currently pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Local Control at 2 years | 2 years
  Local control at 2 years defined as the absence of progression of disease of the treated primary kidney cancer using Responsive Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
Progression-free and Overall survival | week 4-6 post-SBRT, and months: 3,6,9,12,18,24 and 36
  Will be assessed from treatment completion until the date of first progression or date of death from any cause, whichever comes first.
Quality of life of Participants | Baseline, week 4-6 post-SBRT, and months: 3,6,9,12,18,24 and 36
  The Quality of Life will be measured using The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 15 Palliative Care (QLQ-C15-PAL), European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) in renal cell carcinoma patients and The EuroQol 5 Dimension 5 Level (EQ-5D-5L). Each question is scored from 1-4, 1 being the better outcome and 4 being the worst outcome.
Health utilities | Baseline, week 4-6 post-SBRT, and months: 3,6,9,12,18,24 and 36
  Health utilities will be measured using The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 15 Palliative Care (QLQ-C15-PAL), European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) in renal cell carcinoma patients and The EuroQol 5 Dimension 5 Level (EQ-5D-5L). Each question is scored from 1-4, 1 being the better outcome and 4 being the worst outcome.
Late treatment-related toxicities | week 4-6 post-SBRT, and months: 3,6,9,12,18,24 and 36
  Incidence of late treatment related toxicities; assessment made based on the National Cancer Institute Common Toxicity Criteria Adverse Events (NCI CTCAE), version 4.

OTHER OUTCOMES:
Dosimetric parameters | Baseline, Day 3, week 4-6 post-SBRT, and months: 3,6,9,12,18,24 and 36
  Dosimetric parameters (i.e. amount of radiation) to organs at risk (stomach, duodenum, small bowel, large bowel, liver, and normal kidneys) will be collected prospectively for all patients for any correlation between the amount of radiation to specific organs and the presence of toxicities (e.g. stomach upset, nausea/vomiting, diarrhea).
Anatomic Parameters | Baseline and months: 3,6,12,18,24 and 36
  Size, volume and localisation of the kidney tumour relative to organs at risk (stomach, duodenum, liver, normal kidney) will be collected prospectively for all patients.

CONTACTS AND LOCATIONS:
Overall Officials: William Chu, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Center

IPD SHARING:
Plan to Share IPD: No